CLINICAL TRIAL: NCT02311478
Title: (TRIBE) Tracking IUD Bleeding Experiences: An Evaluation of Bleeding Profiles in New Intrauterine Device Users
Brief Title: Tracking IUD Bleeding Experiences: An Evaluation of Bleeding Profiles in New Intrauterine Device Users
Acronym: TRIBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Turok, MD, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 75363
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Intrauterine Devices, Copper; Metrorrhagia; Menstruation; Menstrual Cycle
MeSH Terms: conditions — Metrorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- T380A Copper IUD (Experimental): All participants will receive a T380A copper intrauterine device when enrolled. They can continue using the device for as long as they wish. The study will be completed when 6 months of prospective bleeding data has been collected.
  Interventions: Device: T380A Intrauterine Copper Contraceptive

INTERVENTIONS:
Device: T380A Intrauterine Copper Contraceptive — The T380A is intrauterine device (IUD) that used to prevent pregnancy. It is a soft, flexible T-shaped device made primarily of plastic and copper that is inserted into the uterus.
  Other Names: Paragard

SUMMARY:
This study aims to use validated tools as well as new technology to examine changes in bleeding patterns among women who are initiating the copper T380A IUD.

DETAILED DESCRIPTION:
New users of the intrauterine device (IUD) are most likely to discontinue use within the first six months after insertion. The most common reason for discontinuation of the copper IUD is symptoms related to bleeding. Research looking at disturbances in bleeding patterns among new IUD users is sparse and dated. Perceived changes in vaginal bleeding may impact method satisfaction, acceptability, and continuation. There is a need for updated research evaluating changes in bleeding patterns in order for providers to better counsel patients on what to expect during the months after initiation of an IUD.

A variety of methods to evaluate bleeding profiles are available. The World Health Organization (WHO) published recommendations for methods of collection and analysis of bleeding patterns. The WHO method includes data collection on bleeding days (days when blood loss requires the use of a menstrual pad or tampon) and spotting days (when no protection was needed) using 90-day referent periods. A second tool, the pictorial blood loss assessment chart (PBAC) has been shown to be an inexpensive and objective method of assessing blood loss. The PBAC takes into consideration how heavy blood flow is as well as the number of sanitary napkins and tampons used. Additionally, new technologies (including mobile period tracking applications) have made retrospective collection of bleeding data more feasible and prospective data collection more accurate.

This study aims to incorporate these validated tools as well as new technology to examine changes in bleeding patterns among women who are initiating the copper T380A IUD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women ages 18-40 years with regular, normal menses (lasting between 3-7 days) and who are initiating an IUD
* Women who can provide bleeding information for 3 cycles off of any hormonal contraception (or non-hormonal IUD) and are willing to track bleeding for 180 days
* Women who are between 6 and 12 months postpartum (if they have had normal menses the last 3 cycles)

Exclusion Criteria:

* Use of any hormonal contraceptive method in the previous 3 months
* Irregular duration of menstrual cycles in the last 3 cycles (<21 or >35 days)
* Recent history of menstrual bleeding lasting less than 3 days or greater than 7 days based on self report of the last 3 cycles
* Contraindication to use of the ParaGard® T380A IUD
* Mucopurulent cervicitis at the time of IUD insertion
* Unable to speak, read, and write in English
* Currently pregnant
* Plans for or desire for pregnancy in the next 6 months
* Currently breastfeeding
* Women who are <6 months postpartum
* Participation in any clinical investigation utilizing an investigational drug or medical device or requiring invasive gynecologic procedures within the 30 days prior to enrollment
* Wilson's disease
* Known coagulopathy or bleeding disorder

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2014-12; Primary Completion 2016-08 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, Principal Investigator — Unviersity of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- T380A Copper IUD: All participants will receive a T380A copper intrauterine device when enrolled. The T380A is intrauterine device (IUD) that used to prevent pregnancy. It is a soft, flexible T-shaped device made primarily of plastic and copper that is inserted into the uterus. They can continue using the device for as long as they wish. The study will be completed when 6 months of prospective bleeding data has been collected.
Period: Overall Study
Arm/Group | T380A Copper IUD
Started | 79
IUD Insertion | 78
Completed | 72
Not Completed | 7
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 5
Not completed — Failed IUD Insertion | 1

BASELINE CHARACTERISTICS:
Arm/Group | T380A Copper IUD
Number analyzed (Participants) | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 78
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 66
  Hispanic | 7
  South Pacific Islander | 5
  Black/African American | 2
  Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 78

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Changes in Bleeding Duration Among Women Initiating the Copper T380 IUD During the 90 Days Prior to Initiation Compared to Two 90 Periods After IUD Insertion.
Description: Evaluate bleeding duration among women initiating the copper T380 IUD during the 90 days prior to initiation compared to two 90 periods after IUD insertion. Women will track bleeding after the insertion of the T380A IUD for 180 days. Participants will be contacted monthly to collect data.
Time Frame: 3 months prior to insertion, month 1-month 3 , month 4-month 6
Population: Healthy Women ages 18-40 with menstrual cycle lengths between 21 and 35 days and menses lasting 3 to 7 days, and completed follow up were eligible for participation and analysis. Women were excluded if they reported use of any hormonal contraception in the previous 3 months.
Measure: Mean (95% Confidence Interval); unit: days of bleeding
Arm/Group | T380A Copper IUD
Number analyzed (Participants) | 72
days of bleeding
  3 months prior to insertion | 4.5 [4.1 to 4.9]
  month 1-month3 | 6.0 [5.7 to 6.5]
  month 4-month 6 | 5.5 [5.1 to 5.9]
Statistical Analysis 1: Comparison: T380A Copper IUD; The null hypothesis is that there is no difference between the number of days of bleeding per month at baseline and the days of bleeding per month during 90 days after insertion, and months or 91-180 days following insertion; Test type: Other — Given that this is a observational cohort design we do not use either non-inferiority or equivalence analysis. Using ANOVA we test for differences in the number of days per month of bleeding between the 90 days pre-insertion, the 90 days following insertion, and 91-180 days following insertion; p < 0.05, ANOVA — The p-value is not adjusted for multiple comparisons; df=2; Mean Difference (Net) = 1.77, 95% CI 2-sided [1.2 to 2.3], Standard Error of Mean 0.28
Statistical Analysis 2: Comparison: T380A Copper IUD; The estimation parameter compares the 90 days following to the 90 days prior; Test type: Equivalence — α of 0.05 or lower; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.93, 95% CI 2-sided [0.36 to 1.5]

2. Secondary Outcome: Assess the Relationship of Menstrual Cycle Changes Among Women Initiating the Copper T380 IUD to Method Satisfaction and Continuation at 6 Months Post Insertion.
Description: Determine rates of continuation and level of satisfaction with the IUD during the first 6 months of use.
Time Frame: 6-month post insertion
Measure: Number; unit: percent of patients
Arm/Group | T380A Copper IUD
Number analyzed (Participants) | 78
percent of patients
  satisfied | 51.6
  continuing | 6.4

3. Secondary Outcome: Assess the Relationship of Menstrual Cycle Changes Among Women Initiating the Copper T380 IUD to Sexual Functioning and Satisfaction
Description: % of individuals reporting that their new method had neutral or positive impact of their new contraceptive on their sex life across time points.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | T380A Copper IUD
Number analyzed (Participants) | 72
percentage of participants | 80

ADVERSE EVENTS:
Arm/Group | T380A Copper IUD
All-Cause Mortality (participants affected / at risk) | 0/78
Serious Adverse Events (participants affected / at risk) | 0/78
Other Adverse Events (participants affected / at risk) | 0/78

LIMITATIONS AND CAVEATS:
Limitations

• Baseline bleeding collected retrospectively

Strengths:

* Prospective follow-up with 90% completion
* Uses validated bleeding measures & electronic period trackers to improve reporting accuracy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No